CLINICAL TRIAL: NCT05288101
Title: Effect of Oral Nutritional Supplementation Combined With Impedance Vectors for Dry Weight Adjustment on the Nutritional Status, Hydration Status and Quality of Life in Patients on Chronic Hemodialysis: a Pilot Study
Brief Title: Effect of Oral Nutritional Supplementation Combined With Impedance Vectors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Autonoma de Queretaro (Other)
Collaborators: Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran (Other); Indiana University School of Medicine (Other); Ball State University (Other)
Responsible Party: Principal Investigator, Iris del Carmen Nieves Anaya, Principal Investigator, Universidad Autonoma de Queretaro
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: UAQ-ISSSTE-INCMNSZ-4423632676
Record Dates: First submitted 2021-12-13; First posted 2022-03-18 (Actual); Last update posted 2022-03-18 (Actual); Status verified 2022-03

CONDITIONS: Chronic Kidney Disease Requiring Chronic Dialysis; Overhydration; Undernutrition
Keywords: Dry weight; Undernutrition; Bioelectrical vector analysis; Oral nutrition supplementation; Quality of life
MeSH Terms: conditions — Water Intoxication; Malnutrition

STUDY DESIGN:
Intervention Model Description: Thirty-two chronic HD patients were included in a 6-month randomized pilot study. Patients in SUPL group received a simultaneous intervention consisting of a personalized diet, 245 mL/d ONS and dry weight adjustment through BIVA. Patients in CON group received a personalized diet and dry weight adjustment by BIVA. Anthropometrical, biochemical, dietary, QoL, handgrip strength (HGS) and bioimpedance measurements were performed. Malnutrition Inflammation Score (MIS) was applied.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Control (Active Comparator): Patients in CON group received a personalized diet and dry weight adjustment by BIVA. Anthropometrical, biochemical, dietary, QoL, handgrip strength (HGS) and bioimpedance measurements were performed. Malnutrition Inflammation Score (MIS) was applied
  Interventions: Procedure: Dry weight adjustment through BIVA
- Supplemented (Experimental): Patients in SUPL group received a simultaneous intervention consisting of a personalized diet, 245 mL/d ONS and dry weight adjustment through BIVA, Anthropometrical, biochemical, dietary, QoL, handgrip strength (HGS) and bioimpedance measurements were performed. Malnutrition Inflammation Score (MIS) was applied
  Interventions: Dietary Supplement: Proteinex and Enterex DBT Victus Laboratories; Procedure: Dry weight adjustment through BIVA

INTERVENTIONS:
Dietary Supplement: Proteinex and Enterex DBT Victus Laboratories — The supplement was provided five days per week. Three days a week, the supplement was given at the beginning of the HD session and the patients were instructed to consume it slowly during the next 3 hours. The remaining two days, the supplement was consumed at home and instructed to be consumed between meals. The ONS consisted of one can of polymeric formula (Enterex DBT, Victus Laboratories) and 5.6 g of a protein powder supplement (Proteinex, Victus Laboratories). The final mixture provided 240 kcal, 17 g protein, 8.1 g lipids, 25 g carbohydrates, 4 g dietary fiber, 201 mg sodium, 490 mg calcium, 356 mg phosphorus and 371 mg potassium
  Arms: Supplemented
Procedure: Dry weight adjustment through BIVA — Those participants with post-dialysis vectors located within the 50 or 75% ellipses, were considered to be in dry weight, so they did not require any fluid removal adjustment. However, participants with vectors outside the 75% ellipse were considered overhydrated or dehydrated and dry weight was adjusted. In these patients, if the vectors fell outside the 75% ellipse but within the 95%, above or below the major axis, the established dry weight was adjusted by 0.5 Kg. If the vectors fell outside the 95% ellipse, the weight was adjusted by 1.0 Kg.

SUMMARY:
The objective of this study was to assess the effect of oral nutritional supplementation (ONS) combined with bioelectrical vector analysis (BIVA) on the nutritional and hydration status and the quality of life (QoL) in hemodialysis (HD) patients. Design and Methods: Thirty-two chronic HD patients were included in a 6-month randomized pilot study. Patients in SUPL group received a simultaneous intervention consisting of a personalized diet, 245 mL/d ONS and dry weight adjustment through BIVA. Patients in CON group received a personalized diet and dry weight adjustment by BIVA. Anthropometrical, biochemical, dietary, QoL, handgrip strength (HGS) and bioimpedance measurements were performed. Malnutrition Inflammation Score (MIS) was applied.

DETAILED DESCRIPTION:
This was a randomized, controlled, pilot study. Due to the type of study, no sample size was calculated because the aim was to include all patients available . Patients were randomly assigned to one of two treatments: 1) simultaneous intervention of dry weight adjustment through BIVA, a personalized diet, and 245 mL/d of ONS (SUPL), or 2) dry weight adjustment by BIVA and a personalized diet (CON). Both treatments were given for six months All measurements were made in accordance with good clinical practice and the recommendations of the Helsinki Declaration on human studies. The protocol was registered and approved by the Ethics Committee of the Faculty of Natural Science of the Autonomous University of Queretaro (No. 252FCN2016) and by the Ethics Committee of the ISSSTE in Queretaro. All patients provided written informed consent to participate in this study.

The supplement was provided five days per week. Three days a week, the supplement was given at the beginning of the HD session and the patients were instructed to consume it slowly during the next 3 hours. The remaining two days, the supplement was consumed at home and instructed to be consumed between meals.

The ONS consisted of one can of polymeric formula (Enterex DBT, Victus Laboratories) and 5.6 g of a protein powder supplement (Proteinex, Victus Laboratories). The final mixture provided 240 kcal, 17 g protein, 8.1 g lipids, 25 g carbohydrates, 4 g dietary fiber, 201 mg sodium, 490 mg calcium, 356 mg phosphorus and 371 mg potassium. When the ONS was provided at the HD unit, the mixture was prepared at the hospital´s enteral mixing center and delivered to the patient in a plastic cup with lid and a straw. For the two remaining days, the patients were instructed about the mixture preparation and they were given two cans of supplement and two sealed plastic bags with 5.6 grams of protein powder each one. Adherence to supplement intake was determined by recording the number of servings consumed weekly. For this purpose, at the end of each HD session, the plastic cups were collected to ensure the total consumption of the supplement and for the ONS consumed at home, the patients were asked to return empty cans and plastic bags to the research staff.

Both groups received the intervention to adjust dry weight in order to reach normohydration. Those participants with post-dialysis vectors located within the 50 or 75% ellipses, were considered to be in dry weight, so they did not require any fluid removal adjustment. However, participants with vectors outside the 75% ellipse were considered overhydrated or dehydrated and dry weight was adjusted. In these patients, if the vectors fell outside the 75% ellipse but within the 95%, above or below the major axis, the established dry weight was adjusted by 0.5 Kg. If the vectors fell outside the 95% ellipse, the weight was adjusted by 1.0 Kg.

Patients in both groups also received a personalized diet according to the recommendations of the KDOQI guidelines and the European best practice guidelines on nutrition: 35 Kcal /ideal body weight/day, 1.2 g protein/ideal body weight/day, Na <2000 mg/day, potassium <2000 mg/day, and P <1000 mg/day. Diets were planned and designed by trained renal dietitians and were given to the patients at the beginning of the study. To specify the adequate portion size, food models and photographs of utensils were used. Evaluation of food intake was performed monthly by a three-day food record in order to assess adherence.

ELIGIBILITY:
Inclusion Criteria:

* Patients on chronic HD undergoing thrice weekly hemodialysis (at least three hours per treatment) for more than three months were included.

Exclusion Criteria:

* Patients with amputations of any limb, metal implants, diagnosis of dementia, or current consumption of nutritional supplements were excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2017-06-30 (Actual); Study Completion 2017-06-30 (Actual)

PRIMARY OUTCOMES:
Change in nutritional status from baseline to 6 months | At the beginning of the study (baseline) and at the end of the intervention (six months after starting the intervention).
  Nutritional status was assessed by the Malnutrition Inflammation Score (MIS). MIS is a 27 points maximum scale. According to the total score obtained, the following diagnoses were considered: normal nutritional status (0 points), mild undernutrition (1 - 9 points), moderate undernutrition (10 - 19 points) and severe undernutrition (> 20 points)
Change in hydration status from baseline to 6 months | Every week through study completion (six months).
  Hydration status was evaluated by bioelectrical impedance vector analysis (BIVA). BIA was measured immediately before the start and ten minutes after the end of the mid-week HD session, by the same trained personnel. Individual resistance and reactance values were standardized by the height of each patient (R/H, Xc/H) and then plotted on the reference ellipses of the Mexican population.
  Dehydration was considered when the vector was at the top, outside the 75% ellipses Overhydration was considered when the vector was at the bottom, outside the 75% ellipses Normohydration was considered when the vector was within the ellipses of 50 and 75%

SECONDARY OUTCOMES:
Change in Quality of life evaluation (KDQOL SF) from baseline to 6 months | At the beginning of the study (baseline) and at the end of the intervention (six months after starting the intervention).
  QoL was assessed using the Kidney Disease Quality of Life-Short Form (KDQOL-SF). The instrument includes 36 items. Responses were scored from 0 to 100 points, <50 points meant poor QoL. The higher the score (>50 points), the better QoL.
Change in hand grip strength (HGS) from baseline to 6 months | At the beginning of the study (baseline) and at the end of the intervention (six months after starting the intervention)
  HGS was measured with a dynamometer on the non-fistula side after the HD session, three consecutive times, with a rest period of 1 minute between measurements and the highest value was recorded. Poor strength of the hand and forearm muscles were considered with <20 Kg and <30 Kg for women and men, respectively.
Monthly change in gastrointestinal symptoms evaluation (GSQ) from baseline to 6 months | Every month through study completion (six months).
  Gastrointestinal symptoms were assessed with the self-administered GI symptoms questionnaire (GSQ). The GSQ includes 8 items: anorexia, nausea, vomiting, heartburn, bloating, abdominal pain, constipation and diarrhea. Each symptom is rated between 1 to 5 points, and the higher the score, the more severe the symptoms
Monthly change in calorie intake from baseline to 6 months | Every month through study completion (six months).
  Calorie intake was evaluated by a three-day food record. Patients were asked to record all foods consumed during three days in the same week (one dialysis day, one non-dialysis day, and one weekend day).Three-day food records were analyzed using a nutrient software program and reported as calories consumed per kilogram of weight
Monthly change in protein intake from baseline to 6 months | Every month through study completion (six months).
  Protein intake was evaluated by a three-day food record. Patients were asked to record all foods consumed during three days in the same week (one dialysis day, one non-dialysis day, and one weekend day).Three-day food records were analyzed using a nutrient software program and reported as grams of protein consumed per kilogram of weight
Change in postdialysis weight from baseline to 6 months | Three times a week in every hemodialysis session through study completion (six months).
  Body weight was measured before and after all hemodialysis sessions during the six months of the intervention and reported in kilograms, according to the International Society for the Advancement of Kinanthropometry (ISAK) guidelines.
Change in postdialysis body mass index from baseline to 6 months | Every month through study completion (six months).
  Body mass index was calculated by dividing weight by height squared and reported as kilogram/meters2.
Change in arm muscle circumference from baseline to 6 months | At the beginning of the study (baseline) and at the end of the intervention (six months after starting the intervention)
  Arm circumference and triceps skinfold (TSF) were measured at the end of the mid-week HD session according to the International Society for the Advancement of Kinanthropometry (ISAK) guidelines in triplicate by the same standardized dietitian.
  Arm circumference was calculated usig the following formula: arm circumference (mm) - (3.1416 x triceps skinfold (mm)) and reported in mm
Change in fasting glucose from baseline to 6 months | At the beginning of the study (baseline) and at the end of the intervention (six months after starting the intervention)
  Fasting blood samples were drawn from the vascular access of each participant before the start of the HD session. All tests were performed at the hospital´s clinical laboratory using certified methods.
  Fasting glucose was determined by electric impedance and fluorescence and reported in mg/dl
Change in fasting urea from baseline to 6 months | At the beginning of the study (baseline) and at the end of the intervention (six months after starting the intervention)
  Fasting blood samples were drawn from the vascular access of each participant before the start of the HD session. All tests were performed at the hospital´s clinical laboratory using certified methods.
  Fasting urea was determined by electric impedance and fluorescence and reported in mg/dl
Change in fasting creatinine from baseline to 6 months | At the beginning of the study (baseline) and at the end of the intervention (six months after starting the intervention)
  Fasting blood samples were drawn from the vascular access of each participant before the start of the HD session. All tests were performed at the hospital´s clinical laboratory using certified methods.
  Fasting creatinine was determined by electric impedance and fluorescence and reported in mg/dl
Change in fasting phosphorus from baseline to 6 months | At the beginning of the study (baseline) and at the end of the intervention (six months after starting the intervention)
  Fasting blood samples were drawn from the vascular access of each participant before the start of the HD session. All tests were performed at the hospital´s clinical laboratory using certified methods.
  Fasting phosphorus was determined by electric impedance and fluorescence and reported in mg/dl
Change in fasting sodium from baseline to 6 months | At the beginning of the study (baseline) and at the end of the intervention (six months after starting the intervention)
  Fasting blood samples were drawn from the vascular access of each participant before the start of the HD session. All tests were performed at the hospital´s clinical laboratory using certified methods.
  Fasting sodium was determined by electric impedance and fluorescence and reported in mEq/L
Change in fasting potassium from baseline to 6 months | At the beginning of the study (baseline) and at the end of the intervention (six months after starting the intervention)
  Fasting blood samples were drawn from the vascular access of each participant before the start of the HD session. All tests were performed at the hospital´s clinical laboratory using certified methods.
  Fasting potassium was determined by electric impedance and fluorescence and reported in mEq/L
Change in fasting calcium from baseline to 6 months | At the beginning of the study (baseline) and at the end of the intervention (six months after starting the intervention)
  Fasting blood samples were drawn from the vascular access of each participant before the start of the HD session. All tests were performed at the hospital´s clinical laboratory using certified methods.
  Fasting calcium was determined by electric impedance and fluorescence and reported in mg/dL
Change in fasting albumin from baseline to 6 months | At the beginning of the study (baseline) and at the end of the intervention (six months after starting the intervention)
  Fasting blood samples were drawn from the vascular access of each participant before the start of the HD session. All tests were performed at the hospital´s clinical laboratory using certified methods.
  Fasting albumin was determined by electric impedance and fluorescence and reported in g/dL
Change in fasting transferrin from baseline to 6 months | At the beginning of the study (baseline) and at the end of the intervention (six months after starting the intervention)
  Fasting blood samples were drawn from the vascular access of each participant before the start of the HD session. All tests were performed at the hospital´s clinical laboratory using certified methods.
  Fasting transferrin was determined by chemiluminescence and reported in mg/dL
Change in fasting high-sensitivity C reactive protein from baseline to 6 months | At the beginning of the study (baseline) and at the end of the intervention (six months after starting the intervention)
  Fasting blood samples were drawn from the vascular access of each participant before the start of the HD session. All tests were performed at the hospital´s clinical laboratory using certified methods.
  Fasting high-sensitivity C reactive protein was determined by plate agglutination and reported in mg/dL

CONTACTS AND LOCATIONS:
Overall Officials: Ximena Atilano-Carsi, PhD, Study Director — Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran
Locations (1):
- HD unit of the Social Security Institute for Government Employees (ISSSTE as per initials in Spanish, Querétaro, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nieves-Anaya I, Vargas MB, Mayorga H, Garcia OP, Colin-Ramirez E, Atilano-Carsi X. Comparison of nutritional and hydration status in patients undergoing twice and thrice-weekly hemodialysis: a silent drama in developing countries. Int Urol Nephrol. 2021 Mar;53(3):571-581. doi: 10.1007/s11255-020-02697-3. Epub 2021 Jan 4. PMID 33394280
- [Result] Ikizler TA, Cano NJ, Franch H, Fouque D, Himmelfarb J, Kalantar-Zadeh K, Kuhlmann MK, Stenvinkel P, TerWee P, Teta D, Wang AY, Wanner C; International Society of Renal Nutrition and Metabolism. Prevention and treatment of protein energy wasting in chronic kidney disease patients: a consensus statement by the International Society of Renal Nutrition and Metabolism. Kidney Int. 2013 Dec;84(6):1096-107. doi: 10.1038/ki.2013.147. Epub 2013 May 22. PMID 23698226
- [Result] Hanna RM, Ghobry L, Wassef O, Rhee CM, Kalantar-Zadeh K. A Practical Approach to Nutrition, Protein-Energy Wasting, Sarcopenia, and Cachexia in Patients with Chronic Kidney Disease. Blood Purif. 2020;49(1-2):202-211. doi: 10.1159/000504240. Epub 2019 Dec 18. PMID 31851983
- [Result] Kalantar-Zadeh K, Ikizler TA, Block G, Avram MM, Kopple JD. Malnutrition-inflammation complex syndrome in dialysis patients: causes and consequences. Am J Kidney Dis. 2003 Nov;42(5):864-81. doi: 10.1016/j.ajkd.2003.07.016. PMID 14582032
- [Result] Carrero JJ, Thomas F, Nagy K, Arogundade F, Avesani CM, Chan M, Chmielewski M, Cordeiro AC, Espinosa-Cuevas A, Fiaccadori E, Guebre-Egziabher F, Hand RK, Hung AM, Ikizler TA, Johansson LR, Kalantar-Zadeh K, Karupaiah T, Lindholm B, Marckmann P, Mafra D, Parekh RS, Park J, Russo S, Saxena A, Sezer S, Teta D, Ter Wee PM, Verseput C, Wang AYM, Xu H, Lu Y, Molnar MZ, Kovesdy CP. Global Prevalence of Protein-Energy Wasting in Kidney Disease: A Meta-analysis of Contemporary Observational Studies From the International Society of Renal Nutrition and Metabolism. J Ren Nutr. 2018 Nov;28(6):380-392. doi: 10.1053/j.jrn.2018.08.006. PMID 30348259
- [Result] Sabatino A, Regolisti G, Karupaiah T, Sahathevan S, Sadu Singh BK, Khor BH, Salhab N, Karavetian M, Cupisti A, Fiaccadori E. Protein-energy wasting and nutritional supplementation in patients with end-stage renal disease on hemodialysis. Clin Nutr. 2017 Jun;36(3):663-671. doi: 10.1016/j.clnu.2016.06.007. Epub 2016 Jun 18. PMID 27371993
- [Result] Pupim LB, Majchrzak KM, Flakoll PJ, Ikizler TA. Intradialytic oral nutrition improves protein homeostasis in chronic hemodialysis patients with deranged nutritional status. J Am Soc Nephrol. 2006 Nov;17(11):3149-57. doi: 10.1681/ASN.2006040413. Epub 2006 Oct 4. PMID 17021267
- [Result] Atilano-Carsi X, Miguel JL, Martinez Ara J, Sanchez Villanueva R, Gonzalez Garcia E, Selgas Gutierrez R. [Bioimpedance vector analysis as a tool for the determination and adjustment of dry weight in patients undergoing hemodialysis]. Nutr Hosp. 2015 May 1;31(5):2220-9. doi: 10.3305/nh.2015.31.5.8649. Spanish. PMID 25929397